CLINICAL TRIAL: NCT00999934
Title: Neural Mechanisms Engaged in Control of Eye Movements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: eyemovements01
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-04

CONDITIONS: Degenerative Diseases of the Central Nervous System; Ocular-motor and Vestibular Diseases
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of eye movements is to ensure clear, optimal vision. In order to see clearly, images must be held steady on the retina. Best visual acuity is achieved when the image of the object of interest is brought to and held on the fovea of the retina. Two main types of eye movements are responsible for that: those that keep images stable on the retina (gaze holding mechanisms) and those that change the line of sight (gaze shifting mechanisms). Several functional classes of eye movements have been defined; each has distinctive physiological properties that suit best to its particular task. Thus, vestibular and optokinetic eye movements hold images of the seen world steady on the retina during perturbations of the head. Saccades are rapid eye movements that bring the image of an object of interest, detected in the periphery of vision, onto the fovea where it can be seen best. Smooth pursuit eye movements place the images of a moving target close to fovea. Vergence eye movements place the images of a single object simultaneously onto both foveae.

Each functional class of eye movements relies on a different neural substrate. The clinical significance of it is that impairment of a specific class of eye movement points to involvement of distinct structures or pathways within the brain. Thus, abnormalities of ocular motility are often the clue to the anatomical localization of neurological disorders.

Significance: This study will contribute to understand how the brain governs production of eye movements, and provide better insight on interaction between sensory (visual) and motor (eye movement) system, i.e. sensory-motor interaction. It will also contribute to identify pathophysiological mechanisms underlying human diseases and will improve the investigators' ability to diagnose and encourage development of new therapeutic strategies.

Methods: The investigators will measure eye and head movements using the magnetic scleral search coil technique. The magnetic search coil technique is the most sensitive and accurate technique used in modern ocular motor and vestibular research for measuring horizontal, vertical and torsional eye movements. The coils are easy to apply and well tolerated over a wearing period of up to 45 minutes per recording session.

Population: A grand total of about 250 individuals (normal subjects and patients) will be recruited for the study. Patients will be recruited from the in- and out-patients of the Neurology and Neuro-ophthalmology services of Meir Medical Center. Healthy normal subjects will be recruited from faculty and staff of Meir Medical Center.

Criteria for inclusion/exclusion: The investigators will study patients with neurological disorders causing abnormal eye movements: Degenerative CNS diseases, extrapyramidal disorders, Spino-cerebellar ataxias, Cerebrovascular diseases, demyelinating diseases, Ocular motor and vestibular palsies, Mitochondrial and other ocular myopathies. Only patients who are medically stable and are able to give informed consent will be included in the study. Criteria for excluding subjects will include eye disease such as corneal or scleral abrasion or disease, glaucoma, refractive errors greater than 2 diopters and concurrent medication with CNS-active agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative CNS diseases, extrapyramidal disorders, Spino-cerebellar ataxias, Cerebrovascular diseases, demyelinating diseases, Ocular motor and vestibular palsies, Mitochondrial and other ocular myopathies.
* Patients who are medically stable and are able to give informed consent will be included in the study.

Exclusion Criteria:

* Subjects with eye disease such as corneal or scleral abrasion or disease, glaucoma, refractive errors greater than 2 diopters.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population: A grand total of about 250 individuals (normal subjects and patients) will be recruited for the study. Patients will be recruited from the in- and out-patients of the Neurology and Neuro-ophthalmology services of Meir Medical Center. Healthy normal subjects will be recruited from faculty and staff of Meir Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-07; Primary Completion 2017-06 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Quantitative measure of eye movement and vestibulo-ocular abnormalities | December 1, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Gordon, M.D.; D.Sc., Principal Investigator — Department of Neurology, Meir Medical Center, Kfar Saba and Sackler Faculty of Medicine, Tel Aviv, Israel.
Locations (1):
- Department of Neurology, Kfar Saba, Kfar Saba, Israel